CLINICAL TRIAL: NCT01287247
Title: Prospective, Observational Trial Evaluating Xeomin®(incobotulinumtoxinA) for Cervical Dystonia or Blepharospasm in the United States
Brief Title: Trial Evaluating Xeomin® (incobotulinumtoxinA) for Cervical Dystonia or Blepharospasm in the United States
Acronym: XCiDaBLE
Status: Completed | Type: Observational
Sponsor: Merz North America, Inc. (Industry)
Collaborators: Registrat-Mapi (Other)
Responsible Party: Sponsor
Other Study IDs: MRZ 60201-4066-5
Record Dates: First submitted 2011-01-28; First posted 2011-02-01 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Cervical Dystonia; Blepharospasm
Keywords: Cervical dystonia; Blepharospasm
MeSH Terms: conditions — Torticollis; Blepharospasm | interventions — incobotulinumtoxinA; Botulinum Toxins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cervical Dystonia: The target populations for which the sample size calculations are based are adult subjects aged ≥ 18 years with clinical diagnoses of cervical dystonia.
  Interventions: Biological: Xeomin®
- Blepharospasm: The target populations for which the sample size calculations are based are adult subjects aged ≥ 18 years with clinical diagnoses of blepharospasm.
  Interventions: Biological: Xeomin®

INTERVENTIONS:
Biological: Xeomin® — Xeomin® (incobotulinumtoxinA) at a dose determined by the physician based upon his/her clinical experience with botulinum toxin.
  Other Names: incobotulinumtoxinA; botulinum toxin

SUMMARY:
This is a prospective, observational trial evaluating the "real world" use of Xeomin®(incobotulinumtoxinA). Physicians may enroll patients who are eligible to be treated with a botulinum toxin for cervical dystonia or blepharospasm based upon their clinical experience. The physician must have chosen to treat the patient with Xeomin® (incobotulinumtoxinA) prior to and independent of enrollment in this study. Physicians may choose to treat their subjects with up to 2 treatment cycles (approximately 6 months/subject) of Xeomin® (incobotulinumtoxinA) at a dose determined by the physician based upon his/her clinical experience with botulinum toxin. According and dependent on clinical practice, the investigators expect that subjects will be seen by the investigator for an average of 3 visits (two treatment cycles).

DETAILED DESCRIPTION:
The primary objective of this trial is to collect, evaluate, and report observational data about the clinical use of Xeomin® in a "real world" setting to determine which muscles are injected, the dose used, and how doctors administer the injection.

The secondary objectives of this trial are: To collect and evaluate information about the efficacy of Xeomin®. To collect and evaluate information about the effect of Xeomin® on work productivity and quality of life. To monitor for any serious side effects and non-serious related side effects of Xeomin®

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 years of age or older.
* The physician must have chosen to treat the patient with Xeomin® (incobotulinumtoxinA) prior to and independent of enrollment in this study.
* Subjects who are eligible to be treated with a botulinum toxin for cervical dystonia or blepharospasm based upon the physicians' clinical experience. There are no restrictive subject entry criteria.
* Subjects who are able to read, speak and understand English.

Exclusion Criteria:

* Subjects who are enrolled in any clinical trial (currently or within the past 3 months) in which treatments are imposed by a protocol are not eligible for this trial.
* Any subject for whom botulinum toxin treatment would be contraindicated; see Xeomin® Prescribing Information for further details.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects 18 years of age or older. The physician must have chosen to treat the patient with Xeomin® (incobotulinumtoxinA) prior to and independent of enrollment in this study.
Sampling Method: Probability Sample
Enrollment: 688 (Actual)
Dates: Start 2011-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Determination of injection patterns and techniques | Two treatment cycles (approximately 6 months/subject)
  To collect, evaluate and report observational data about the clinical use of Xeomin® in a "real world" setting to determine injection patterns and use of guidance techniques.

SECONDARY OUTCOMES:
To collect and evaluate efficacy of Xeomin®(incobotulinumtoxinA) including onset and offset of effect as well as improvement of disease specific and global illness severity | Two treatment cycles (approximately 6 months/subject)

CONTACTS AND LOCATIONS:
Overall Officials: Hubert H. Fernandez, MD, FAAN, Principal Investigator — Center for Neurological Restoration
Locations (70):
- United States (70):
  - Site #001052, Cullman, Alabama
  - Scottsdale, Arizona
  - Site # 001974, Tucson, Arizona
  - Site #001046, Encinitas, California
  - Site # 001822, Fountain Valley, California
  - Site # 001852, La Jolla, California
  - Merz Investigative Site #001986, Los Angeles, California
  - Site # 001924, Los Gatos, California
  - Site # 001005, Newport Beach, California
  - Site # 001973, Sacramento, California
  - Site # 001977, New Haven, Connecticut
  - Site # 001901, Washington D.C., District of Columbia
  - Site # 001803, Boca Raton, Florida
  - Site # 001805, North Palm Beach, Florida
  - Site # 001955, Sarasota, Florida
  - Site # 001823, St. Petersburg, Florida
  - Site # 001972, Chicago, Illinois
  - Site #001057, Glenview, Illinois
  - Site #001978, Lake Bluff, Illinois
  - Site # 001820, Winfield, Illinois
  - Site # 001995, Munster, Indiana
  - Site # 001833, Overland Park, Kansas
  - Site # 001047, Baton Rouge, Louisiana
  - Site # 001849, Baltimore, Maryland
  - Site # 001053, Boston, Massachusetts
  - Site # 001816, Roseville, Michigan
  - Site # 001848, Warren, Michigan
  - Site # 001028, Bloomington, Minnesota
  - Site # 001834, Eagan, Minnesota
  - Site # 001957, Minneapolis, Minnesota
  - Site # 001802, Des Peres, Missouri
  - Site # 001838, St Louis, Missouri
  - Site # 001010, Las Vegas, Nevada
  - Site # 001954, Reno, Nevada
  - Site #001961, Toms River, New Jersey
  - Site # 001860, Kingston, New York
  - Site # 001041, New York, New York
  - Site # 001921, New York, New York
  - Site # 001910, New York, New York
  - Site # 001034, North Syracuse, New York
  - Site # 001013, Syracuse, New York
  - Site # 001951, Durham, North Carolina
  - Merz Investigative Site # 001840, Bellevue, Ohio
  - Site # 001812, Cleveland, Ohio
  - Site # 001826, Columbus, Ohio
  - Site # 001815, Tulsa, Oklahoma
  - Site # 001916, Bend, Oregon
  - Site # 001839, Medford, Oregon
  - Site #001000, Collegeville, Pennsylvania
  - Site # 001959, Philadelphia, Pennsylvania
  - Site #001032, Wynnewood, Pennsylvania
  - Site # 001893, Spartanburg, South Carolina
  - Site # 001922, Chattanooga, Tennessee
  - Site # 001889, Columbia, Tennessee
  - Site # 001831, Memphis, Tennessee
  - Site # 001836, Nashville, Tennessee
  - Merz Investigative Site # 001055, Bedford, Texas
  - Site # 001055, Bedford, Texas
  - Site # 001037, Bedford, Texas
  - Site # 001817, Dallas, Texas
  - Site # 001809, Dallas, Texas
  - Site # 001022, Houston, Texas
  - Site # 001813, Houston, Texas
  - Site #001802, Houston, Texas
  - Site # 001960, Tyler, Texas
  - Site # 001962, Alexandria, Virginia
  - Site # 001980, Fishersville, Virginia
  - Site #001979, Virginia Beach, Virginia
  - Site # 001881, Kirkland, Washington
  - Site # 001800, Spokane, Washington